CLINICAL TRIAL: NCT06735586
Title: The Effect of Hip Strengthening Exercises and Taping on Pain, Function and Balance in Patients With Patellofemoral Pain Syndrome With Dynamic Valgus
Brief Title: The Effect of Hip Strengthening Exercises and Taping in Patients With PFP With Dynamic Valgus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Dilber Karagozoglu Coskunsu, Assoc. Prof., Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BahcesehirUn; Dilber Karagözoğlu Coşkunsu (Other: Bahcesehir University)
Record Dates: First submitted 2023-04-08; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Patellofemoral Pain; Valgus Deformity
Keywords: Dynamic Knee Valgus; Patellofemoral Pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Intervention Model Description: By randomly dividing the individuals investigators included in our study into two groups, investigators applied only the hip and quadriceps strengthening program to one group and the additional Mulligan rigid taping technique to the hip and quadriceps strengthening exercises in the other group, and examined the first and post-test measurements investigators will make before and after each group separately, at the same time. İnvestigators are planning to evaluate the results investigators have obtained by making comparisons between groups in both groups. Dilber Coşkunsu, who is a blind evaluator, will make the evaluations. The person making the evaluation will make an evaluation without knowing which treatment the patient is receiving.
Who Masked: Outcomes Assessor
Masking Description: Outcome measuements were performed by blind assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular control exercises plus taping (Experimental): İnvestigators will apply the Mulligan knee taping technique to the participants in the randomized exercise and taping group, in addition to the hip focused and quadriceps strengthening exercises, 3 times a week for a total of 6 weeks.
  Interventions: Procedure: neuromuscular control exercise and taping
- Neuromuscular control exercises (Active Comparator): All of the 17 participants participating in the study will be included in the 6-week exercise program investigators created after the initial evaluations. Exercises will be done 3 times a week, 10 sets of each exercise. And the participants will be given a rest period of 3 minutes between each set.
  Interventions: Procedure: neuromuscular control exercise

INTERVENTIONS:
Procedure: neuromuscular control exercise — All of the 17 participants participating in the study will be included in the 6-week exercise program investigators created after the initial evaluations. Exercises will be done 3 times a week, 10 sets of each exercise. And the participants will be given a rest period of 3 minutes between each set.1st and 2nd (5 times) week exercise program: Non-weight bearing exercises will be given in the first week; lateral hip abduction, clam shell exercises, and bridging exercises. 3rd and 4th week (5 times) exercises: This week investigators will give controlled weight lifting exercises:pelvic drop exercise, single leg squat exercise,step down exercise,single leg raise exercise. 4th and 5 th week exercise: lateral band walks, side lunges, forward lunges, and back lunges. 5 th and 6 th week exercise: Plyometric exercises: jump exercise, BOSU single knee scales exercise,resistive single leg squats,resisting vertical bridge.
  Arms: Neuromuscular control exercises
Procedure: neuromuscular control exercise and taping — Exercises and taping will be done 3 times a week, 10 sets of each exercise. Mulligan Knee Taping Application: The application was made with Protape 38mm x 10 m rigid tape. The application will be performed in the participant's foot, with the hip and knee in internal rotation, and the knee in 20º flexion. The tape will be applied starting from the head of the fibula, passing over the tibia anteriorly, passing under the medial joint line of the knee and ending at the back of the knee, bringing the tibia to internal rotation.
  Arms: Neuromuscular control exercises plus taping

SUMMARY:
The aim of the study is to investigate the effects of isolated quadriceps and hip strengthening exercises and both strengthening exercises and mulligan knee taping technique on pain, functional level and balance in patients with dynamic knee valgus and patellofemoral pain. In addition, in the groups investigators will create as randomized controlled, investigators give only strengthening exercise to one group and apply both exercise and taping to the other group and to investigate whether Mulligan taping, which is applied in addition to exercise in the treatment, has an effect on valgus correction, pain, functional level and balance, and contributes to the literature. It will also become clear how effective the strengthening exercises will be in correcting the dynamic valgus, how much participants will reduce patellofemoral pain, and whether they have an effect on the functional level and balance. There are not enough studies in the literature on strengthening exercises in patients with patellofemoral pain with dynamic valgus. İnvestigators will contribute to the literature by evaluating the effect of hip and quadriceps strengthening exercises on dynamic knee valgus and patellofemoral pain with 2D video analysis method and evaluating the results concretely. In addition to the strengthening exercises that investigators will apply to the other group, our other research target is to evaluate the Mulligan knee taping technique with 2D video analysis method and to investigate whether Mulligan knee taping treatment has an effect on the correction of dynamic valgus.

DETAILED DESCRIPTION:
A total of 34 patients with anterior knee pain and dynamic valgus will be included in the study and randomly divided into 2 groups as Exercise and Taping (n=17) and Exercise (n=17). Hip and quadriceps strengthening exercises will be applied to the patients in the exercise group 3 times a week for a total of 6 weeks, and both strengthening exercises and mulligan rigid knee taping will be applied to the patients in the Exercise and Taping group, again for 6 weeks and 3 times a week. If the participants in the study have bilateral anterior knee pain, the more symptomatic side will be included in the study.

Outcome measurements will be performed on the baseline (first day-before first treatment) and at the end of the 6 weeks treatment program.

NCSS (Number Cruncher Statistical System) 2007 (Kaysville, Utah,USA) program will be used for statistical analysis. While evaluating the study data, descriptive statistical methods (Mean, Standard Deviation, Median, Frequency, Ratio, Minimum, Maximum) as well as the distribution of the data will be evaluated with the Shapiro-Wilk Test.

Mann-Whitney U Test will be used in comparisons of two groups that cannot show normal distribution of quantitative data, and Student's t test will be used in case of normal distribution. Significance will be evaluated at the p<0.05 level.

ELIGIBILITY:
Inclusion Criteria:

* Anterior knee pain lasting more than 2 months
* > 10 degrees frontal plane valgus angle
* At least 3 pains on the 10 cm VAS scale in the last week
* Have symptoms for at least 2 months
* Patients aged 18 to 50 years
* To have at least 2 of the pains that occur during squatting, climbing stairs, descending and sitting

Exclusion Criteria:

* Neurological disease or sequelae
* Having an orthopedic injury that may affect lower extremity kinematics
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-04-02 (Actual)

PRIMARY OUTCOMES:
Anterior knee pain scale | 6 week
  measures the index function. the lowest 0 takes the highest 100 value.

SECONDARY OUTCOMES:
Visual analog scale | 6 week
  İnvestigators will evaluate pain with the VAS scale.The lowest value will be scored as 0 and the highest value as 10.Those with a value of 3 or more will be included in the study. The first and last day will be evaluated.
Y Balance Test | 6 week
  Dynamic balance measurements of patients will be evaluated with Y balance test. In the test set up, 3 measuring tapes will be glued to the ground with an angle of 120 between them. The patient will be asked to stand on one foot at the intersection of these 3 tapes, reach with the tip of the toe in these 3 directions with the other foot, anterior, posteromedial and posterolateral, and return to the starting position.
Frontal plane projection angle | 6 week
  In our study, our participants will be evaluated with single leg squat test and 2D video analysis method on the first and last day.Individuals will be asked to stand on one leg and bend their knees. The dynamic knee valgus of the participants who are positioned in 45º-60º flexion and observed from the frontal plane for 5 seconds will be evaluated.
Patellar tilt test | 6 week
  It is used to assess the tension of the lateral retinacular structures. With the patient lying in the supine position with the knee fully extended, investigators will evaluate with 2 fingers or 4 fingers whether there is a difference between the medial and lateral vertical heights of the patella. A lateral tilt is considered positive if the lateral side height is less than the medial side height.
Muscle strength measurement | 6 week
  Muscle strength measurements will be made with MicroFET2 hand dynamometer, whose reliability has been proven as isometric muscle strength measurement. Knee extension, hip external rotation, hip extension, hip abduction muscle strength will be measured.
Hip external rotation and internal rotation E.H.A measurements | 6 week
  The patient is sitting with his legs hanging off the table from the knee, and the measurement will be made with a goniometer.
Q angle measurement | 6 week
  The q angle is the angle between the line extending from the anterior superior of the spina iliaca to the midpoint of the patella and the line extending from the midpoint of the patella to the tuberositas tibia while the patient is standing.

CONTACTS AND LOCATIONS:
Locations (1):
- BahcesehirUni, Istanbul, Beşiktaş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No